CLINICAL TRIAL: NCT03619083
Title: Assessment of Sensory Gating, Attention, and Executive Control in Breast Cancer
Status: Active, not recruiting | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: The City College of New York (Other)
Responsible Party: Sponsor
Other Study IDs: 18-240
Record Dates: First submitted 2018-07-17; First posted 2018-08-07 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2025-02

CONDITIONS: Breast Cancer
Keywords: Assessments; Sensory Gating; Attention; Executive Control; 18-240
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Breast cancer patients treated with chemotherapy
  Interventions: Other: SAE battery; Behavioral: Assessments
- patients not exposed to chemotherapy
  Interventions: Other: SAE battery; Behavioral: Assessments
- healthy controls
  Interventions: Other: SAE battery; Behavioral: Assessments

INTERVENTIONS:
Other: SAE battery — The SAE battery yields 12 variables.
  Other Names: Sensory-Attention-Executive
Behavioral: Assessments — Assessments of their neurocognitive performance will be assessed longitudinally, at 4 time points: prior to adjuvant treatment (post-surgery); 1 month (with a +4 week window) post-chemotherapy; and again at the 12 and 24 months (with a +4 week window) post-treatment time points. These assessment time points are denoted as T1 though T4, respectively. The assessment schedule for the HC and CT- groups will be yoked against that of the CT+ cohort.

SUMMARY:
This study is being done to find out if a new series of evaluations called the SAE (Sensory-Attention-Executive) Battery can help researchers learn more about how cancer treatment does or does not change the way the brain processes/filters information, emotions, attention span, and behavior by comparing the results of the SAE Battery with traditional evaluations like questionnaires.

ELIGIBILITY:
Inclusion Criteria:

For Patients:

* As per medical record or self-report, female
* As per medical record or self-report, age 40-75 at diagnosis of a new primary histological confirmed adenocarcinoma breast cancer
* As per medical record or self-report, AJCC stages 0-3 breast cancer
* As per medical record or self-report, post-surgery for current breast cancer diagnosis (surgery includes cryosurgery/cryotherapy)
* Score of < 11 on the Blessed Orientation-Memory-Concentration Test (BOMC)
* As per medical record or self-report, if currently taking psychoactive medications (excluding gabapentin and including but not limited to antidepressants and anxiolytics) on a daily basis, dose must have been stable at least two months prior to enrollment.
* English fluent (as per self-report, fluency of "well" or "very well", and having a reasonable comprehension of the study conversation in the opinion of the research staff)**

For Healthy Controls:

* As per medical record or self-report, female
* As per medical record or self-report, age 40-75
* As per medical record or self-report, if currently taking psychoactive medications (including but not limited to antidepressants and anxiolytics), dose must have been stable at least two months prior to enrollment.
* As per self report, no history of cancer except non-melanoma/basal cell skin cancer/squamous cell skin carcinoma and, at the discretion of the PI, early stage secondary cancer diagnoses treated only with surgery
* Score of < 11 on the Blessed Orientation-Memory-Concentration Test (BOMC)
* English fluent (as per self-report, fluency of "well" or "very well", and having a reasonable comprehension of the study conversation in the opinion of the research staff)**

Exclusion Criteria:

For All Participants:

* As per medical record or self-report, diagnosis of neurodegenerative disorder that affects cognitive function (e.g. Alzheimer's disease, Parkinson's disease, Multiple Sclerosis, Dementia, Seizure Disorders, etc.)
* As per medical record or self report, history of stroke or head injury resulting in a structural lesion on neuropsych imaging, persistent cognitive difficulties impacting work or daily life, or required cognitive rehabilitation
* As per medical record or self report, a diagnosis of a Schizophrenia Spectrum Disorder, substance use disorder, Bipolar Disorder or Schizotypal personality disorder. Schizophrenia Spectrum Disorders include Schizophrenia, Schizophreniform disorder, Schizoaffective disorder, Delusional disorder, Brief psychotic disorder, and Attenuated Psychotic Disorder.
* As per medical record or self-report, visual or auditory impairment that would preclude ability to complete the assessments (e.g. history of significant macular degeneration or being unable to correct hearing with hearing aides)
* As per medical record or self-report, use of methotrexate (Amethopterin, Rhematrex, Trexall) or rituximab (Rituxin) for rheumatoid arthritis, psoriasis or Crohn's disease, or cyclophosphamide (Cytoxan, Neosar) for Lupus.
* As per medical record or self-report, history of treatment using radiation, chemotherapy, and/or Tamoxifen or Aromatase-inhibitors

For Patients only:

* As per medical record or self-report, history of another type of cancer or prior breast cancer diagnosis except non-melanoma/basal cell skin cancer/squamous cell skin carcinoma and, at the discretion of the PI, early stage secondary cancer diagnoses treated only with surgery
* As per medical record or self-report, disease recurrence. ** Language verification: For both patients and controls, prior to enrollment, all will be asked the following two questions by an RSA to verify English fluency necessary for participation in the study:

  1. How well do you speak English? (must respond "Well" or "Very well" when given the choices of Very well, Well, Not well, Not at all, Don't know, or Refused)
  2. What is your preferred language for healthcare? (must respond English)

Ages: 40 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Breast cancer
Study Population: A total of 300 participants (n = 100 breast cancer patients treated with chemotherapy, n = 100 breast cancer patients without chemotherapy treatment, n = 100 matched controls).
Sampling Method: Non-Probability Sample
Enrollment: 187 (Actual)
Dates: Start 2018-07-13 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
congnitive changes in patients | 3 years
  using the Sensory-Attention-Executive Battery

CONTACTS AND LOCATIONS:
Overall Officials: James Root, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm